CLINICAL TRIAL: NCT00578500
Title: Study That Establishes the Potential of Fertility Preservation in Young Female Patients by Oocyte in Vitro Maturation and Cryopreservation and Ovarian Cortex Cryopreservation and Transplantation
Brief Title: Fertility Preservation by Ovarian and Oocyte Cryopreservation
Acronym: HFPP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Ariel Revel, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2819; 29-18/1/08
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2002-01

CONDITIONS: Female Patients Aged 5-35 Prior to Systemic Chemotherapy; With Significant Risk of Ovarian Toxicity
Keywords: chemotherapy, female, fertility preservation, gonadotoxicity; oophorectomy, in vitro maturation, ovarian cryopreservation,; oocyte cryopreservation, ovarian transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OCCT (Active Comparator): Patients referred to ovarian cryopreservation.
  Interventions: Procedure: ovarian transplantation

INTERVENTIONS:
Procedure: ovarian transplantation — Patients will undergo laparoscopic oophorectomy, aspiration of oocytes and maturation followed by cryopreservation. In case of ovarian failure and approval by treating physicians, restoration of fertility will be attempted by thawing of oocytes or by transplantation of ovarian cortex to induce ovulation and obtain oocytes for fertilization and embryo transfer.

SUMMARY:
Success rates of cancer treatment have increased significantly resulting in many girls and young women who are treated now and will be cancer survivors. Nevertheless, cancer treatment may result in long term side effects. Damage to the ovaries may result in serious difficulty to become pregnant in the future. The risk of this happening depends, among others upon patient's age, disease and type of treatment she undergoes. Medical research is continuously looking into ways to preserve female fertility by using less toxic protocols. Yet, keeping your eggs outside the body during treatment is an interesting option which as is routine for boys preserving sperm before cancer treatment. This research attempts to freeze eggs either in the ovarian tissue or individually.

DETAILED DESCRIPTION:
Advances in early detection and increasing success of chemotherapy have made cancer therapy a curable disease. In children and adolescents with cancer, cure rates approach 75%. These cure rates are achieved in great part due to the use of intensive chemotherapy, and in some cases, radiation. The use of these treatment modalities is associated with significant toxicity, including the potential for gonadal damage and subsequent reduced fertility. Aggressive chemotherapy is, however, usually gonadotoxic and results in infertility in many pediatric patients. Ovarian damage is drug and dose dependant and increases with patient age at treatment. Increasing numbers of young cancer survivors are therefore experiencing infertility related to their past cancer treatment. Having children thus becomes an important issue for young cancer patients.

Cryopreservation of sperm is an effective method that is offered to pre- and post-adolescent males. Female gametes were however, not readily amenable to cryopreservation though the use of vitrification recently resulted in improved results. Nevertheless, this method is not applicable for young girls as it requires prolonged induction of ovulation and vaginal sonography to complete aspiration of oocytes. Similarly, In vitro fertilization (IVF) may be offered only to patients beyond adolescence. Ovulation induction requires a few weeks delay in the initiation of cancer treatment.

Since ovarian stimulation is generally not a feasible option for young girls and adolescents, strategies for preserving fertility in these patients usually include ovarian cryopreservation, an experimental technology with some success in animal studies, recently resulting in few deliveries following human transplantations. Although the technique remains investigational, it is being increasingly offered to women undergoing cancer treatment. In prepubertal girls ovarian cryopreservation is the only option for potentially preserving ovarian function. As we and others have shown, it is probable that methods of ovarian transplantation with vascular anastomosis will be applied in the future.

We have recently recommended that following individual consultation by a multi-disciplinary team, all female pediatric cancer patients and their families should be counseled regarding side effects of chemotherapy and be offered ovarian preservation.

The methodology of ovarian cortex preservation, pioneered by Gosden is currently routine in many centers in a few countries. Nevertheless, it is realized that the future use of this cryopreserved ovarian cortex may be limited due to cellular injury during cryopreservation and due to the tissue ischemic damage following transplantation.

Furthermore, cryobanking of ovarian cortex preserves only the smallest (primordial and primary) follicles, since all preovulatory antral follicles, which contain GV stage oocytes will not survive the procedure. We thus currently propose to all patients undergoing ovarian cryopreservation to perform integrated oocyte aspiration from antral follicles of the tissue, followed by in vitro maturation (IVM) and oocyte cryopreservation as an additional fertility-preserving method. The aim of this study was to analyze oocyte detection and IVM success rates in young girls and adolescents using this combined method.

ELIGIBILITY:
Inclusion Criteria:

* patients before chemotherapy with significant risk to future fertility

Exclusion Criteria:

* high operative risk

Ages: 5 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2000-01; Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
risks involved in laparoscopic oophorectomy | 10 years

SECONDARY OUTCOMES:
Ability to restore fertility by ovarian cortex transplantation | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Revel, MD, Principal Investigator — Hadassah university hospital
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel

REFERENCES:
- [Result] Revel A, Koler M, Simon A, Lewin A, Laufer N, Safran A. Oocyte collection during cryopreservation of the ovarian cortex. Fertil Steril. 2003 May;79(5):1237-9. doi: 10.1016/s0015-0282(02)04963-4. No abstract available. PMID 12738527